CLINICAL TRIAL: NCT05437939
Title: Identifying Opportunities for Prevention of Adverse Outcomes Following Female Genital
Brief Title: Adverse Outcomes Following Female Genital Fistula Repair
Acronym: Mulisa
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Infectious Diseases Research Collaboration, Uganda (Other); Makerere University (Other)
Responsible Party: Sponsor
Other Study IDs: A137001; R01HD101570 (NIH)
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Female Genital Fistula; Incontinence
Keywords: Surgical repair breakdown; Obstetrics fistula; Fistula; Incontinence; Urine incontinence; Fistula repair; Fistula recurrence
MeSH Terms: conditions — Fistula; Nocturnal Enuresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Following genital fistula repair, fistula repair breakdown and recurrence, persistent and incidence incontinence are major adverse outcomes, limiting women's health and wellbeing. Using a prospective design, the investigators seek to identify modifiable risk factors to establish key targets for intervention, followed by qualitative work to refine the feasibility and acceptability of potential intervention strategies.

DETAILED DESCRIPTION:
Although improved global surgical access has begun to reduce the significant physical, psychosocial, and economic consequences of fistula, women with successful surgery face adverse post-repair risks. Emerging research has identified post-repair fistula recurrence in up to 14% of women following surgery, with many recurrences occurring within the first 12 months. Post-repair incontinence continues in up to 33% of women despite closed fistula, with some women developing incident incontinence after previously successful resolution through fistula surgery. However, the limited evidence base on factors contributing to adverse outcomes limits interventions to improve women's health and quality of life following genital fistula repair.

The investigators hypothesize that important independent predictors of vesicovaginal fistula repair breakdown and recurrence will include indications of fistula severity, strenuous labor, early resumption of sexual intercourse and subsequent pregnancy. Further modifiable characteristics whose potential contribution the investigators seek to establish for these adverse outcomes include other post-repair behaviors and exposures. To test these hypotheses and explore additional contributors to adverse outcomes, the investigators will leverage the research infrastructure the investigators have developed at several fistula repair sites in Uganda to lead a 3-year longitudinal cohort study of up to 1000 women following genital fistula repair. The investigators will collect data on sociodemographic characteristics, fistula and repair-related characteristics at fistula repair, and data on post-repair behaviors and exposures quarterly. If participants report key symptoms (recurrence and incontinence), the investigators will confirm these outcomes by clinical validation through physical examination. The investigators will calculate incidence and establish temporal relationships of a range of exposures with adverse outcomes to identify key targets for intervention. The investigators will then engage key stakeholders in iterative qualitative work framed by key behavioral and implementation science theories to enhance translation of our quantitative findings into intervention strategies that are feasible and acceptable in this context. This mixed-methods work has a strong potential to directly influence programming to reduce adverse outcomes following genital fistula repair.

Aim 1: Identify predictors of post-repair fistula breakdown and recurrence. The investigators will use survival analysis methods to compare baseline and time-varying patient characteristics of women in our longitudinal cohort who develop post-repair fistula breakdown and recurrence compared to those who do not. Assessment will focus on mutable factors fistula repair-related characteristics and post-repair behaviors and exposures, accounting for immutable participant baseline sociodemographic and fistula characteristics.

Aim 2: Identify predictors and characteristics of post-repair incontinence. Specifically, the investigators seek to identify predictors of post-repair incontinence (see Aim 1) in our longitudinal cohort, focusing on: a) persistent incontinence following surgery at multiple time-points; and b) time to incident incontinence among women whose incontinence was initially resolved by surgery; using similar methods to Aim 1.

Aim 3: Identify feasible and acceptable strategies for modifying key risk factors of adverse outcome. To improve the translation of our research findings from Aims 1 and 2 into practice, the investigators will engage in an iterative process with key stakeholders to understand their perspectives on potential strategies for modifying important risk factors influencing post-repair fistula breakdown, recurrence, and incontinence. The investigators will purposively recruit a sub-sample of cohort participants (n=40) and other key stakeholders such as families, community members, and fistula care providers (n=40) for in-depth interview, followed by iterative participatory work with our qualitative sample to refine acceptability and feasibility concerns and ultimately to guide intervention strategy development.

ELIGIBILITY:
Inclusion Criteria:

* Vesicovaginal fistula
* Completed surgery with confirmed surgical closure
* Age 15 or above, with ages 15-17 meeting criteria for emancipated minor
* Capable of providing informed consent

Exclusion Criteria:

* None beyond above

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to n=1000 women with successful (closed) vesicovaginal fistula repair who are 18 and older or 15-17 year old emancipated minors (per Ugandan law) will be eligible to participate from fistula surgery centers and hospitals participating in the study as recruitment sites.
Sampling Method: Non-Probability Sample
Enrollment: 802 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Time to post-repair fistula breakdown | Through 36 months following study enrollment
  Proportion of women who experience fistula breakdown (a reopening of the fistula following repair, prior to the complete healing or de novo fistula occurrence as confirmed by a positive methylene blue dye test) and reported as the incidence by the total person-time observed and measured up to 36 months following index fistula repair
Time to post-repair urinary incontinence | Through 36 months following study enrollment
  Proportion of women who experience post-repair incontinence (as measured through urinary incontinence with confirmed negative methylene blue dye test indicated complete fistula closure) measured up to 36 months following index fistula repair

CONTACTS AND LOCATIONS:
Overall Officials: Alison El Ayadi, ScD, Principal Investigator — University of California, San Francisco
Locations (1):
- Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Bernis L. Obstetric fistula: guiding principles for clinical management and programme development, a new WHO guideline. Int J Gynaecol Obstet. 2007 Nov;99 Suppl 1:S117-21. doi: 10.1016/j.ijgo.2007.06.032. Epub 2007 Sep 18. PMID 17880979
- [Background] Wall LL, Arrowsmith SD, Briggs ND, Browning A, Lassey A. The obstetric vesicovaginal fistula in the developing world. Obstet Gynecol Surv. 2005 Jul;60(7 Suppl 1):S3-S51. doi: 10.1097/00006254-200507001-00002. No abstract available. PMID 16034313
- [Background] Hilton P. Vesico-vaginal fistulas in developing countries. Int J Gynaecol Obstet. 2003 Sep;82(3):285-95. doi: 10.1016/s0020-7292(03)00222-4. PMID 14499975
- [Background] Hilton P, Ward A. Epidemiological and surgical aspects of urogenital fistulae: a review of 25 years' experience in southeast Nigeria. Int Urogynecol J Pelvic Floor Dysfunct. 1998;9(4):189-94. doi: 10.1007/BF01901602. PMID 9795822
- [Background] Arrowsmith S, Hamlin EC, Wall LL. Obstructed labor injury complex: obstetric fistula formation and the multifaceted morbidity of maternal birth trauma in the developing world. Obstet Gynecol Surv. 1996 Sep;51(9):568-74. doi: 10.1097/00006254-199609000-00024. PMID 8873157
- [Background] Wall LL, Arrowsmith SD, Briggs ND, Lassey A. Urinary Incontinence in the Developing World: The Obstetric Fistula. In: Abrams P, Cardozo L, Khoury S, Wein A, eds. Incontinence. Plymouth, U.K.: Health Publication Ltd; 2002.
- [Background] Zeleke BM, Ayele TA, Woldetsadik MA, Bisetegn TA, Adane AA. Depression among women with obstetric fistula, and pelvic organ prolapse in northwest Ethiopia. BMC Psychiatry. 2013 Sep 26;13:236. doi: 10.1186/1471-244X-13-236. PMID 24070342
- [Background] Browning A, Fentahun W, Goh JT. The impact of surgical treatment on the mental health of women with obstetric fistula. BJOG. 2007 Nov;114(11):1439-41. doi: 10.1111/j.1471-0528.2007.01419.x. Epub 2007 Sep 27. PMID 17903234
- [Background] Goh JT, Sloane KM, Krause HG, Browning A, Akhter S. Mental health screening in women with genital tract fistulae. BJOG. 2005 Sep;112(9):1328-30. doi: 10.1111/j.1471-0528.2005.00712.x. PMID 16101616
- [Background] Browning A. Risk factors for developing residual urinary incontinence after obstetric fistula repair. BJOG. 2006 Apr;113(4):482-5. doi: 10.1111/j.1471-0528.2006.00875.x. Epub 2006 Feb 20. PMID 16489933
- [Background] Nielsen HS, Lindberg L, Nygaard U, Aytenfisu H, Johnston OL, Sorensen B, Rudnicki M, Crangle M, Lawson R, Duffy S. A community-based long-term follow up of women undergoing obstetric fistula repair in rural Ethiopia. BJOG. 2009 Aug;116(9):1258-64. doi: 10.1111/j.1471-0528.2009.02200.x. Epub 2009 May 14. PMID 19459865
- [Background] Delamou A, Utz B, Delvaux T, Beavogui AH, Shahabuddin A, Koivogui A, Leveque A, Zhang WH, De Brouwere V. Pregnancy and childbirth after repair of obstetric fistula in sub-Saharan Africa: Scoping Review. Trop Med Int Health. 2016 Nov;21(11):1348-1365. doi: 10.1111/tmi.12771. Epub 2016 Sep 6. PMID 27596732
- [Background] Delamou A, Delvaux T, El Ayadi AM, Tripathi V, Camara BS, Beavogui AH, Romanzi L, Cole B, Bouedouno P, Diallo M, Barry TH, Camara M, Diallo K, Leveque A, Zhang WH, De Brouwere V. Fistula recurrence, pregnancy, and childbirth following successful closure of female genital fistula in Guinea: a longitudinal study. Lancet Glob Health. 2017 Nov;5(11):e1152-e1160. doi: 10.1016/S2214-109X(17)30366-2. Epub 2017 Sep 21. PMID 28941996
- [Background] Frajzyngier V, Ruminjo J, Barone MA. Factors influencing urinary fistula repair outcomes in developing countries: a systematic review. Am J Obstet Gynecol. 2012 Oct;207(4):248-58. doi: 10.1016/j.ajog.2012.02.006. Epub 2012 Feb 20. PMID 22475385
- [Background] El Ayadi AM, Barageine J, Korn A, Kakaire O, Turan J, Obore S, Byamugisha J, Lester F, Nalubwama H, Mwanje H, Tripathi V, Miller S. Trajectories of women's physical and psychosocial health following obstetric fistula repair in Uganda: a longitudinal study. Trop Med Int Health. 2019 Jan;24(1):53-64. doi: 10.1111/tmi.13178. Epub 2018 Nov 18. PMID 30372572
- [Background] Bengtson AM, Kopp D, Tang JH, Chipungu E, Moyo M, Wilkinson J. Identifying Patients With Vesicovaginal Fistula at High Risk of Urinary Incontinence After Surgery. Obstet Gynecol. 2016 Nov;128(5):945-953. doi: 10.1097/AOG.0000000000001687. PMID 27741181
- [Background] Evoh NJ, Akinla O. Reproductive performance after the repair of obstetric vesico-vaginal fistulae. Ann Clin Res. 1978 Dec;10(6):303-6. PMID 742828
- [Background] Browning A, Menber B. Women with obstetric fistula in Ethiopia: a 6-month follow up after surgical treatment. BJOG. 2008 Nov;115(12):1564-9. doi: 10.1111/j.1471-0528.2008.01900.x. PMID 19035992
- [Background] Kayondo M, Wasswa S, Kabakyenga J, Mukiibi N, Senkungu J, Stenson A, Mukasa P. Predictors and outcome of surgical repair of obstetric fistula at a regional referral hospital, Mbarara, western Uganda. BMC Urol. 2011 Dec 7;11:23. doi: 10.1186/1471-2490-11-23. PMID 22151960
- [Background] Muleta M. Socio-demographic profile and obstetric experience of fistula patients managed at the Addis Ababa Fistula Hospital. Ethiop Med J. 2004 Jan;42(1):9-16. PMID 15884272
- [Background] Wall LL. Obstetric vesicovaginal fistula as an international public-health problem. Lancet. 2006 Sep 30;368(9542):1201-9. doi: 10.1016/S0140-6736(06)69476-2. PMID 17011947
- [Background] Khisa AM, Nyamongo IK. Still living with fistula: an exploratory study of the experience of women with obstetric fistula following corrective surgery in West Pokot, Kenya. Reprod Health Matters. 2012 Dec;20(40):59-66. doi: 10.1016/S0968-8080(12)40661-9. PMID 23245409
- [Background] El Ayadi AM, Barageine JK, Miller S, Byamugisha J, Nalubwama H, Obore S, Korn A, Sukumar S, Kakaire O, Mwanje H, Lester F, Turan JM. Women's experiences of fistula-related stigma in Uganda: a conceptual framework to inform stigma-reduction interventions. Cult Health Sex. 2020 Mar;22(3):352-367. doi: 10.1080/13691058.2019.1600721. Epub 2019 Apr 30. PMID 31035913
- [Background] Baker Z, Bellows B, Bach R, Warren C. Barriers to obstetric fistula treatment in low-income countries: a systematic review. Trop Med Int Health. 2017 Aug;22(8):938-959. doi: 10.1111/tmi.12893. Epub 2017 Jul 20. PMID 28510988
- [Background] Barageine JK, Beyeza-Kashesya J, Byamugisha JK, Tumwesigye NM, Almroth L, Faxelid E. "I am alone and isolated": a qualitative study of experiences of women living with genital fistula in Uganda. BMC Womens Health. 2015 Sep 10;15:73. doi: 10.1186/s12905-015-0232-z. PMID 26359255
- [Background] Mwini-Nyaledzigbor PP, Agana AA, Pilkington FB. Lived experiences of Ghanaian women with obstetric fistula. Health Care Women Int. 2013;34(6):440-60. doi: 10.1080/07399332.2012.755981. PMID 23641897
- [Background] Mselle LT, Moland KM, Evjen-Olsen B, Mvungi A, Kohi TW. "I am nothing": experiences of loss among women suffering from severe birth injuries in Tanzania. BMC Womens Health. 2011 Nov 15;11:49. doi: 10.1186/1472-6874-11-49. PMID 22082132
- [Background] Wilson AL, Chipeta E, Kalilani-Phiri L, Taulo F, Tsui AO. Fertility and pregnancy outcomes among women with obstetric fistula in rural Malawi. Int J Gynaecol Obstet. 2011 Jun;113(3):196-8. doi: 10.1016/j.ijgo.2011.01.006. Epub 2011 Apr 1. PMID 21457981
- [Background] Azhar RA, Bochner B, Catto J, Goh AC, Kelly J, Patel HD, Pruthi RS, Thalmann GN, Desai M. Enhanced Recovery after Urological Surgery: A Contemporary Systematic Review of Outcomes, Key Elements, and Research Needs. Eur Urol. 2016 Jul;70(1):176-187. doi: 10.1016/j.eururo.2016.02.051. Epub 2016 Mar 9. PMID 26970912
- [Background] Korol E, Johnston K, Waser N, Sifakis F, Jafri HS, Lo M, Kyaw MH. A systematic review of risk factors associated with surgical site infections among surgical patients. PLoS One. 2013 Dec 18;8(12):e83743. doi: 10.1371/journal.pone.0083743. eCollection 2013. PMID 24367612
- [Background] Carey MP, Goh JT, Fynes MM, Murray CJ. Stress urinary incontinence after delayed primary closure of genitourinary fistula: a technique for surgical management. Am J Obstet Gynecol. 2002 May;186(5):948-53. doi: 10.1067/mob.2002.122247. PMID 12015520
- [Background] Murray C, Goh JT, Fynes M, Carey MP. Urinary and faecal incontinence following delayed primary repair of obstetric genital fistula. BJOG. 2002 Jul;109(7):828-32. doi: 10.1111/j.1471-0528.2002.00124.x. PMID 12135221
- [Background] Goh JT, Krause H, Tessema AB, Abraha G. Urinary symptoms and urodynamics following obstetric genitourinary fistula repair. Int Urogynecol J. 2013 Jun;24(6):947-51. doi: 10.1007/s00192-012-1948-z. Epub 2012 Oct 25. PMID 23096530
- [Background] Boaz A, Hanney S, Borst R, O'Shea A, Kok M. How to engage stakeholders in research: design principles to support improvement. Health Res Policy Syst. 2018 Jul 11;16(1):60. doi: 10.1186/s12961-018-0337-6. PMID 29996848
- [Background] Jull JE, Davidson L, Dungan R, Nguyen T, Woodward KP, Graham ID. A review and synthesis of frameworks for engagement in health research to identify concepts of knowledge user engagement. BMC Med Res Methodol. 2019 Nov 21;19(1):211. doi: 10.1186/s12874-019-0838-1. PMID 31752691
- [Background] Shelef DQ, Rand C, Streisand R, Horn IB, Yadav K, Stewart L, Foushee N, Waters D, Teach SJ. Using stakeholder engagement to develop a patient-centered pediatric asthma intervention. J Allergy Clin Immunol. 2016 Dec;138(6):1512-1517. doi: 10.1016/j.jaci.2016.10.001. Epub 2016 Oct 12. PMID 27744029
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Birken SA, Powell BJ, Presseau J, Kirk MA, Lorencatto F, Gould NJ, Shea CM, Weiner BJ, Francis JJ, Yu Y, Haines E, Damschroder LJ. Combined use of the Consolidated Framework for Implementation Research (CFIR) and the Theoretical Domains Framework (TDF): a systematic review. Implement Sci. 2017 Jan 5;12(1):2. doi: 10.1186/s13012-016-0534-z. PMID 28057049
- [Background] Bentley MR, Mitchell N, Sutton L, Backhouse SH. Sports nutritionists' perspectives on enablers and barriers to nutritional adherence in high performance sport: A qualitative analysis informed by the COM-B model and theoretical domains framework. J Sports Sci. 2019 Sep;37(18):2075-2085. doi: 10.1080/02640414.2019.1620989. Epub 2019 May 24. PMID 31124393
- [Background] Chater AM, Williams J, Courtenay M. The prescribing needs of community practitioner nurse prescribers: A qualitative investigation using the theoretical domains framework and COM-B. J Adv Nurs. 2019 Nov;75(11):2952-2968. doi: 10.1111/jan.14170. Epub 2019 Sep 3. PMID 31423627
- [Background] Courtenay M, Rowbotham S, Lim R, Peters S, Yates K, Chater A. Examining influences on antibiotic prescribing by nurse and pharmacist prescribers: a qualitative study using the Theoretical Domains Framework and COM-B. BMJ Open. 2019 Jun 19;9(6):e029177. doi: 10.1136/bmjopen-2019-029177. PMID 31221892
- [Background] Thompson LM, Diaz-Artiga A, Weinstein JR, Handley MA. Designing a behavioral intervention using the COM-B model and the theoretical domains framework to promote gas stove use in rural Guatemala: a formative research study. BMC Public Health. 2018 Feb 14;18(1):253. doi: 10.1186/s12889-018-5138-x. PMID 29444650
- [Background] Flannery C, McHugh S, Anaba AE, Clifford E, O'Riordan M, Kenny LC, McAuliffe FM, Kearney PM, Byrne M. Enablers and barriers to physical activity in overweight and obese pregnant women: an analysis informed by the theoretical domains framework and COM-B model. BMC Pregnancy Childbirth. 2018 May 21;18(1):178. doi: 10.1186/s12884-018-1816-z. PMID 29783933
- [Background] Browning A, Patel TL. FIGO initiative for the prevention and treatment of vaginal fistula. Int J Gynaecol Obstet. 2004 Aug;86(2):317-22. doi: 10.1016/j.ijgo.2004.05.003. No abstract available. PMID 15289120
- [Background] Uganda Bureau of Statistics, ICF. Uganda Demographic and Health Survey 2016. Kampala, Uganda: UBOS and ICF, 2018.
- [Background] Uganda Ministry of Health. National Obstetric Fistula Strategy 2011/2012-2015/2016. Kampala: Uganda Ministry of Health; 2011.
- [Background] Direct Relief. Global Fistula Map. 2013. http://www.globalfistulamap.org/ (accessed Nov 1 2015).
- [Background] McCurdie FK, Moffatt J, Jones K. Vesicovaginal fistula in Uganda. J Obstet Gynaecol. 2018 Aug;38(6):822-827. doi: 10.1080/01443615.2017.1407301. Epub 2018 Mar 9. PMID 29523027
- [Background] Direct Relief, Fistula Foundation. Global Fistula Hub. 2019. https://www.globalfistulahub.org/ (accessed December 1 2020).
- [Background] El Ayadi A, Nalubwama H, Barageine J, Neilands TB, Obore S, Byamugisha J, Kakaire O, Mwanje H, Korn A, Lester F, Miller S. Development and preliminary validation of a post-fistula repair reintegration instrument among Ugandan women. Reprod Health. 2017 Sep 2;14(1):109. doi: 10.1186/s12978-017-0372-8. PMID 28865473
- [Background] DataReportal 2021. Digital 2021 Uganda, 2021.
- [Background] Uganda Communications Commission. Market Performance Report: 1Q21. Kampala, Uganda: Uganda Communications Commission, 2021.
- [Background] Stamatakos M, Sargedi C, Stasinou T, Kontzoglou K. Vesicovaginal fistula: diagnosis and management. Indian J Surg. 2014 Apr;76(2):131-6. doi: 10.1007/s12262-012-0787-y. Epub 2012 Dec 14. PMID 24891778
- [Background] FIGO, Partners. Global Competency-Based Fistula Surgery Trainining Manual; 2011.
- [Background] Hancock B. First Steps In Vesico-Vaginal Fistula Repair. London: The Royal Society of Medicine Press Ltd; 2005.
- [Background] Hancock B, Browning A. A text book of practical obstetric fistula surgery. London: Royal Society of Medicine Press Ltd; 2009.
- [Background] Kees Waaldijk. Step by step surgery of vesico vaginal fistulae. Edinburgh (UK): Campion Press; 1998.
- [Background] Waaldijk K. Obstetrics fistula surgery art and science. Edinburgh, UK: Campion Press; 2008.
- [Background] Wall LL. Preventing obstetric fistulas in low-resource countries: insights from a Haddon matrix. Obstet Gynecol Surv. 2012 Feb;67(2):111-21. doi: 10.1097/OGX.0b013e3182438788. PMID 22325301
- [Background] Jackson S, Donovan J, Brookes S, Eckford S, Swithinbank L, Abrams P. The Bristol Female Lower Urinary Tract Symptoms questionnaire: development and psychometric testing. Br J Urol. 1996 Jun;77(6):805-12. doi: 10.1046/j.1464-410x.1996.00186.x. PMID 8705212
- [Background] Martin F, Russell S, Seeley J. The WHOQOL BREF questionnaire in Luganda: Validation with a sample including people living with HIV in Uganda. Working Paper 46. Norwich, United Kingdom: School of International Development, University of East Anglia, 2013.
- [Background] Webster J, Nicholas C, Velacott C, Cridland N, Fawcett L. Validation of the WHOQOL-BREF among women following childbirth. Aust N Z J Obstet Gynaecol. 2010 Apr;50(2):132-7. doi: 10.1111/j.1479-828X.2009.01131.x. PMID 20522068
- [Background] Lundberg P, Rukundo G, Ashaba S, Thorson A, Allebeck P, Ostergren PO, Cantor-Graae E. Poor mental health and sexual risk behaviours in Uganda: a cross-sectional population-based study. BMC Public Health. 2011 Feb 21;11:125. doi: 10.1186/1471-2458-11-125. PMID 21338500
- [Background] Lundberg P, Cantor-Graae E, Rukundo G, Ashaba S, Ostergren PO. Urbanicity of place of birth and symptoms of psychosis, depression and anxiety in Uganda. Br J Psychiatry. 2009 Aug;195(2):156-62. doi: 10.1192/bjp.bp.108.051953. PMID 19648549
- [Background] Hatcher AM, Tsai AC, Kumbakumba E, Dworkin SL, Hunt PW, Martin JN, Clark G, Bangsberg DR, Weiser SD. Sexual relationship power and depression among HIV-infected women in Rural Uganda. PLoS One. 2012;7(12):e49821. doi: 10.1371/journal.pone.0049821. Epub 2012 Dec 26. PMID 23300519
- [Background] Bolton P, Wilk CM, Ndogoni L. Assessment of depression prevalence in rural Uganda using symptom and function criteria. Soc Psychiatry Psychiatr Epidemiol. 2004 Jun;39(6):442-7. doi: 10.1007/s00127-004-0763-3. PMID 15205728
- [Background] Martin F, Russell S, Seeley J. Toward an understanding of the impact of HIV medication on quality of life in Uganda. 2013 Division of Health Psychology Annual Conference. Brighton, UK; 2013.
- [Background] Rosenberg M. Society and the adolescent self-image. Princeton, NJ: Princeton University Press; 1965.
- [Background] Holzemer WL, Human S, Arudo J, Rosa ME, Hamilton MJ, Corless I, Robinson L, Nicholas PK, Wantland DJ, Moezzi S, Willard S, Kirksey K, Portillo C, Sefcik E, Rivero-Mendez M, Maryland M. Exploring HIV stigma and quality of life for persons living with HIV infection. J Assoc Nurses AIDS Care. 2009 May-Jun;20(3):161-8. doi: 10.1016/j.jana.2009.02.002. PMID 19427593
- [Background] Holzemer WL, Uys L, Makoae L, Stewart A, Phetlhu R, Dlamini PS, Greeff M, Kohi TW, Chirwa M, Cuca Y, Naidoo J. A conceptual model of HIV/AIDS stigma from five African countries. J Adv Nurs. 2007 Jun;58(6):541-51. doi: 10.1111/j.1365-2648.2007.04244.x. Epub 2007 May 1. PMID 17484748
- [Background] Nakigudde J, Musisi S, Ehnvall A, Airaksinen E, Agren H. Adaptation of the multidimensional scale of perceived social support in a Ugandan setting. Afr Health Sci. 2009 Aug 1;9 Suppl 1(Suppl 1):S35-41. PMID 20589159
- [Background] Osman A, Lamis DA, Freedenthal S, Gutierrez PM, McNaughton-Cassill M. The multidimensional scale of perceived social support: analyses of internal reliability, measurement invariance, and correlates across gender. J Pers Assess. 2014;96(1):103-12. doi: 10.1080/00223891.2013.838170. Epub 2013 Oct 3. PMID 24090236
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Cox CM, Hindin MJ, Otupiri E, Larsen-Reindorf R. Understanding couples' relationship quality and contraceptive use in Kumasi, Ghana. Int Perspect Sex Reprod Health. 2013 Dec;39(4):185-94. doi: 10.1363/3918513. PMID 24393724
- [Background] Flynn KE, Lin L, Cyranowski JM, Reeve BB, Reese JB, Jeffery DD, Smith AW, Porter LS, Dombeck CB, Bruner DW, Keefe FJ, Weinfurt KP. Development of the NIH PROMIS (R) Sexual Function and Satisfaction measures in patients with cancer. J Sex Med. 2013 Feb;10 Suppl 1(0 1):43-52. doi: 10.1111/j.1743-6109.2012.02995.x. PMID 23387911
- [Background] LP S. Stata 16 Base Reference Manual. College Station, TX: Stata Press, 2019.
- [Background] Kalbfleisch JD, Prentice RL. The Statistical Analysis of Failure Time Data. 2nd ed. New York: Wiley; 2002.
- [Background] Gutierrez R. Parametric frailty and shared frailty survival models. Stata Journal 2002; 2: 22-44
- [Background] Hernan MA, Robins JM. Estimating causal effects from epidemiological data. J Epidemiol Community Health. 2006 Jul;60(7):578-86. doi: 10.1136/jech.2004.029496. PMID 16790829
- [Background] Austin PC, Stuart EA. Moving towards best practice when using inverse probability of treatment weighting (IPTW) using the propensity score to estimate causal treatment effects in observational studies. Stat Med. 2015 Dec 10;34(28):3661-79. doi: 10.1002/sim.6607. Epub 2015 Aug 3. PMID 26238958
- [Background] Rosenbaum PR. Model-Based Direct Adjustment. Journal of the American Statistical Association 1987; 82(398): 387-94
- [Background] Hirano K, Imbens GW. The propensity score with continuous treatments. In: Gelman A, Meng XL, eds. Applied Bayesian Modeling and Causal Inference from Incomplete-Data Perspectives. West Sussex, England: Wiley; 2004.
- [Background] Strobl C, Malley J, Tutz G. An introduction to recursive partitioning: rationale, application, and characteristics of classification and regression trees, bagging, and random forests. Psychol Methods. 2009 Dec;14(4):323-48. doi: 10.1037/a0016973. PMID 19968396
- [Background] StataCorp LP. Stata Survey Data Reference Manua, Release 14. College Station, Texas, 2015.
- [Background] Keith RE, Crosson JC, O'Malley AS, Cromp D, Taylor EF. Using the Consolidated Framework for Implementation Research (CFIR) to produce actionable findings: a rapid-cycle evaluation approach to improving implementation. Implement Sci. 2017 Feb 10;12(1):15. doi: 10.1186/s13012-017-0550-7. PMID 28187747
- [Background] Saunders B, Sim J, Kingstone T, Baker S, Waterfield J, Bartlam B, Burroughs H, Jinks C. Saturation in qualitative research: exploring its conceptualization and operationalization. Qual Quant. 2018;52(4):1893-1907. doi: 10.1007/s11135-017-0574-8. Epub 2017 Sep 14. PMID 29937585
- [Background] Bernard HR, Ryan GW. Analyzing Qualitative Data: Systematic Approaches. Thousand Oaks, CA: SAGE Publication, Inc. ; 2010.
- [Background] Slinger G, Trautvetter L, Browning A, Rane A. Out of the shadows and 6000 reasons to celebrate: An update from FIGO's fistula surgery training initiative. Int J Gynaecol Obstet. 2018 Jun;141(3):280-283. doi: 10.1002/ijgo.12482. Epub 2018 Apr 10. PMID 29634084
- [Derived] El Ayadi AM, Obore S, Kirya F, Miller S, Korn A, Nalubwama H, Neuhaus J, Getahun M, Eyul P, Twine R, Andrew EVW, Barageine JK. Identifying opportunities for prevention of adverse outcomes following female genital fistula repair: protocol for a mixed-methods study in Uganda. Reprod Health. 2024 Jan 4;21(1):2. doi: 10.1186/s12978-023-01732-7. PMID 38178156
- [Derived] El Ayadi AM, Obore S, Kirya F, Miller S, Korn A, Nalubwama H, Neuhaus J, Getahun M, Eyul P, Twine R, Andrew EVW, Barageine JK. Identifying Opportunities for Prevention of Adverse Outcomes Following Female Genital Fistula Repair: Protocol for a Mixed-Methods Study in Uganda. Res Sq [Preprint]. 2023 May 5:rs.3.rs-2879899. doi: 10.21203/rs.3.rs-2879899/v1. PMID 37205399